CLINICAL TRIAL: NCT00611975
Title: Effect of Serotonin Reuptake Inhibitors on Gonadal Steroid Hormones
Brief Title: Effect of Antidepressants on Sex Hormone Levels and Sexual Functioning
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R21MH071543 (NIH); R21MH071543 (NIH); DNBBS 73-MCR
Record Dates: First submitted 2008-02-06; First posted 2008-02-11 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Gonadal Steroid Hormones; Healthy Volunteers; Antidepressant Side Effects; Fluoxetine; Bupropion; Prolactin; Testosterone; Estradiol; Progesterone; Sexual Function; Serotonin Reuptake Inhibitors; 17-OH Pregnenolone
MeSH Terms: interventions — Fluoxetine; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Participants will receive treatment with fluoxetine for 2 months
  Interventions: Drug: Fluoxetine
- B (Experimental): Participants will receive treatment with bupropion for 2 months
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Fluoxetine — Participants will begin taking 10 mg of fluoxetine, once a day by mouth, on the first day of their second menstrual cycle during the study. Dosage will be increased to 20 mg of fluoxetine once a day after 7 days, to be maintained until the luteal phase (start of ovulation) of menstrual cycle 3. If side effects are intolerable, the dose will be lowered to 10 mg of fluoxetine per day. Participants will undergo a total of 2 months of treatment with fluoxetine.
  Other Names: Prozac, Sarafem
  Arms: A
Drug: Bupropion — Participants will begin taking 150 mg of bupropion, once a day by mouth, on the first day of their second menstrual cycle during the study. Dosage will be increased to 300 mg of bupropion once a day after 7 days, to be maintained until the luteal phase of menstrual cycle 3. If side effects are intolerable, the dose will be decreased to 150 mg of bupropion per day. Participants will undergo a total of 2 months of treatment with bupropion.
  Other Names: Wellbutrin, Zyban
  Arms: B

SUMMARY:
This study will evaluate the effect of antidepressants on sex hormone levels in women and if the potential changes in sex hormone levels are related to sexual side effects.

DETAILED DESCRIPTION:
Depression is a leading cause of disability in women, with women being two times more likely than men to develop depression. Depression affects a person's body, thoughts, mood, and behavior, often making normal day-to-day functioning difficult. Fortunately, depression is a condition that is highly treatable with one or more of the antidepressant medications and forms of psychotherapy available. Serotonin reuptake inhibitors (SRIs) are a recent class of antidepressants that have been successful in alleviating symptoms of depression. Although the side effects of SRIs are less than those of other types of antidepressants, a number of people taking SRIs experience sexual dysfunction, including reduced desire and difficulty with orgasm. It is believed that SRI treatment may interfere with gonadal production of steroid hormones, thus leading to changes in sexual function. This study will compare the effects of the SRI fluoxetine with the effects of the non-SRI bupropion on circulating levels of sex hormones in healthy women and on any related sexual side effects.

Participation in this study will last 3 months. Potential participants will undergo initial screening, which will involve a blood draw, drug and pregnancy tests, physical exam, electrocardiogram, and psychiatric diagnostic interview. Participants will also complete an interview and questionnaire about sexual functioning. All eligible participants will then be asked to return for a total of 9 study visits over 3 months.

Participants will undergo 1 month of baseline hormonal sampling and 2 months of daily treatment with either fluoxetine or bupropion. The study visits will be scheduled around three points in the menstrual cycle (early follicular, ovulatory, and luteal), with each visit including a blood draw and repeat questionnaire on sexual functioning. Participants will be asked to perform daily urine tests, beginning 10 days after the start of menstruation and continuing for up to 8 days until detection of the luteinizing hormone surge, which signals ovulation. Participants will be asked to keep a diary of luteinizing hormone surges, dates of menstruation, and sexual activities. At the Month 3 visit, participants will discontinue their assigned medication and will complete their final blood draw and questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycles that are 25 to 35 days in length during the 1 year prior to study entry
* Willing to engage in sexual activity, alone or with a partner, at least weekly for the duration of the study
* Willing to use effective birth control (e.g., condom, diaphragm with spermicide, tubal ligation, nonhormonal intrauterine device,, partner with vasectomy) for the duration of the study

Exclusion Criteria:

* Medical illness that may contribute to sexual dysfunction or affect steroid hormone levels
* Body mass index (BMI) greater than 30
* Elevated testosterone at screening
* History of seizure disorder
* Consumes more than 10 alcoholic beverages per week

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Altemus, MD, Principal Investigator — Weill Medical College of Cornell University

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoxetine: Participants will receive treatment with fluoxetine for 2 months
  Fluoxetine: Participants will begin taking 10 mg of fluoxetine, once a day by mouth, on the first day of their second menstrual cycle during the study. Dosage will be increased to 20 mg of fluoxetine once a day after 7 days, to be maintained until the luteal phase (start of ovulation) of menstrual cycle 3. If side effects are intolerable, the dose will be lowered to 10 mg of fluoxetine per day. Participants will undergo a total of 2 months of treatment with fluoxetine.
- Bupropion: Participants will receive treatment with bupropion for 2 months
  Bupropion: Participants will begin taking 150 mg of bupropion, once a day by mouth, on the first day of their second menstrual cycle during the study. Dosage will be increased to 300 mg of bupropion once a day after 7 days, to be maintained until the luteal phase of menstrual cycle 3. If side effects are intolerable, the dose will be decreased to 150 mg of bupropion per day. Participants will undergo a total of 2 months of treatment with bupropion.
Period: Overall Study
Arm/Group | Fluoxetine | Bupropion
Started | 45 | 38
Completed | 40 | 30
Not Completed | 5 | 8
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Pregnancy | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine | Bupropion | Total
Number analyzed (Participants) | 45 | 38 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (5.5) | 27.9 (6.4) | 27.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 37 | 32 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 14 | 24
  White | 25 | 18 | 43
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in 17-OH Pregnenolone
Description: Hormone levels at early follicular, ovulation, and luteal phase of 3 menstrual cycles which included baseline, month 1 of daily antidepressant treatment and month 2 of daily antidepressant treatment. Effects of the two antidepressant treatments and menstrual cycle on hormone level were examined.
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: All subjects enrolled were included in the mixed model analysis. For mean results at each timepoint in the data table below, some subjects were not included due to missing blood samples or samples collected outside the specified cycle phase window.
Measure: Mean (Standard Error); unit: ng/dl
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 45 | 38
ng/dl
  Baseline month follicular: number analyzed (Participants) | 44 | 38
  Baseline month follicular | 120 (14) | 158 (17)
  Baseline month ovulation: number analyzed (Participants) | 27 | 20
  Baseline month ovulation | 171 (46) | 170 (23)
  Baseline month luteal | 141 (18) | 189 (22)
  Treatment month 1 follicular: number analyzed (Participants) | 42 | 38
  Treatment month 1 follicular | 151 (15) | 184 (39)
  Treatment month 1 ovulation: number analyzed (Participants) | 24 | 18
  Treatment month 1 ovulation | 122 (20) | 142 (22)
  Treatment month 1 luteal: number analyzed (Participants) | 40 | 30
  Treatment month 1 luteal | 109 (14) | 163 (20)
  Treatment month 2 follicular: number analyzed (Participants) | 40 | 32
  Treatment month 2 follicular | 101 (9) | 138 (19)
  Treatment month 2 ovulation: number analyzed (Participants) | 21 | 14
  Treatment month 2 ovulation | 174 (32) | 176 (20)
  Treatment month 2 luteal: number analyzed (Participants) | 34 | 28
  Treatment month 2 luteal | 167 (32) | 161 (21)
Statistical Analysis 1: Comparison: Fluoxetine vs Bupropion; Blood draws were scheduled for early follicular, ovulatory and luteal phases. Menstrual phase for blood samples were re-assigned to phase based on time to onset of next menstrual period. Early follicular(35-21 days before next menstrual period (NMP)), Ovulatory (16-12 before NMP) luteal (11-3 days before NMP); Test type: Superiority or Other; p > 0.8, Mixed Models Analysis
Statistical Analysis 2: Comparison: Fluoxetine vs Bupropion; This secondary analysis examined main effect of menstrual cycle phase on hormone levels; Test type: Superiority or Other; p > 0.4, Mixed Models Analysis

2. Secondary Outcome: Change in Arizona Sexual Experiences Scale (ASEX)
Description: A five-item scale with each item scored from 1 to 6. Score range is 5 to 30. Higher scores indicate more sexual dysfunction.
  Scores at early follicular, ovulation, and luteal phase of 3 menstrual cycles which included baseline month, month 1 of daily antidepressant treatment and month 2 of daily antidepressant treatment. Differential effects of the two antidepressant treatments and menstrual cycle on ASEX scores were examined.
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: All subjects enrolled were included in the mixed model analysis. For mean results at each timepoint in the data table below, some subjects were not included due to missing questionnaire samples or samples collected outside the specified cycle phase window.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 45 | 38
score on a scale
  Baseline month follicular: number analyzed (Participants) | 40 | 38
  Baseline month follicular | 13.1 (.5) | 12.9 (.7)
  Baseline month ovulation: number analyzed (Participants) | 20 | 19
  Baseline month ovulation | 11.3 (0.6) | 12.1 (1.1)
  Baseline month luteal: number analyzed (Participants) | 41 | 38
  Baseline month luteal | 14.0 (0.8) | 12.4 (0.7)
  Treatment month 1 follicular: number analyzed (Participants) | 45 | 33
  Treatment month 1 follicular | 15.1 (.9) | 13.6 (10.9)
  Treatment month 1 ovulation: number analyzed (Participants) | 24 | 18
  Treatment month 1 ovulation | 15.0 (1.0) | 12.6 (1.0)
  Treatment month 1 luteal: number analyzed (Participants) | 40 | 33
  Treatment month 1 luteal | 14.8 (.7) | 13.8 (0.8)
  Treatment month 2 follicular: number analyzed (Participants) | 40 | 31
  Treatment month 2 follicular | 14.4 (0.7) | 14.3 (0.9)
  Treatment month 2 ovulation: number analyzed (Participants) | 14 | 14
  Treatment month 2 ovulation | 13.6 (1.2) | 15.2 (1.4)
  Treatment month 2 luteal: number analyzed (Participants) | 29 | 25
  Treatment month 2 luteal | 15.1 (0.7) | 14.4 (1.0)
Statistical Analysis 1: Comparison: Fluoxetine vs Bupropion; Asex questionnaires were scheduled for early follicular, ovulatory and luteal phases. Menstrual phase for ASEX scores were re-assigned to phase based on time to onset of next menstrual period. Follicular(35-21 days before next menstrual period (NMP)), Ovulatory (16-12 before NMP) luteal (11-2 days before NMP); Test type: Superiority or Other; p > 0.6, Mixed Models Analysis
Statistical Analysis 2: Comparison: Fluoxetine vs Bupropion; This secondary analysis examined main effect of menstrual cycle phase on ASEX scores; Test type: Superiority or Other; p > 0.6, Mixed Models Analysis

3. Secondary Outcome: Change in Free Testosterone
Description: Free testosterone was calculated from total testosterone ng/ml divided by sex hormone binding globulin (SHBG) nmol/l multiplied by 100. Hormone levels at early follicular, ovulation, and luteal phase of 3 menstrual cycles which included baseline month, month 1 of daily antidepressant treatment and month 2 of daily antidepressant treatment. Differential effects of the two antidepressant treatments and menstrual cycle on hormone levels were examined.
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: as for outcome 1
Measure: Mean (Standard Error); unit: calculated ratio
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 45 | 38
calculated ratio
  Baseline month follicular: number analyzed (Participants) | 44 | 38
  Baseline month follicular | .41 (.03) | .44 (.02)
  Baseline month ovulation: number analyzed (Participants) | 27 | 19
  Baseline month ovulation | .52 (.05) | .69 (.09)
  Baseline month luteal | .47 (.04) | .47 (.04)
  Treatment month 1 follicular: number analyzed (Participants) | 44 | 38
  Treatment month 1 follicular | .39 (.02) | .51 (.04)
  Treatment month 1 ovulation: number analyzed (Participants) | 26 | 16
  Treatment month 1 ovulation | .41 (.04) | .65 (.13)
  Treatment month 1 luteal: number analyzed (Participants) | 43 | 35
  Treatment month 1 luteal | .49 (.04) | .48 (.05)
  Treatment month 2 follicular: number analyzed (Participants) | 40 | 32
  Treatment month 2 follicular | .36 (.03) | .40 (.04)
  Treatment month 2 ovulation: number analyzed (Participants) | 21 | 14
  Treatment month 2 ovulation | .50 (.04) | .81 (.20)
  Treatment month 2 luteal: number analyzed (Participants) | 39 | 28
  Treatment month 2 luteal | .50 (.07) | .44 (.06)
Statistical Analysis 1: Comparison: Fluoxetine vs Bupropion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .01, Mixed Models Analysis
Statistical Analysis 2: Comparison: Fluoxetine vs Bupropion; This secondary analysis examined main effect of menstrual cycle phase on hormone levels; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis

4. Secondary Outcome: Change in Estradiol
Description: Hormone levels at early follicular, ovulation, and luteal phase of 3 menstrual cycles which included baseline, month 1 of daily antidepressant treatment and month 2 of daily antidepressant treatment. Effects of the two antidepressant treatments and menstrual cycle on hormone levels were examined.
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 45 | 38
pg/ml
  Baseline month follicular: number analyzed (Participants) | 42 | 38
  Baseline month follicular | 42 (5) | 38 (3)
  Baseline month ovulation: number analyzed (Participants) | 26 | 19
  Baseline month ovulation | 131 (14) | 134 (20)
  Baseline Month Luteal | 107 (7) | 109 (8)
  Treatment month 1 follicular: number analyzed (Participants) | 41 | 37
  Treatment month 1 follicular | 41 (5) | 42 (6)
  Treatment month 1 ovulation: number analyzed (Participants) | 24 | 17
  Treatment month 1 ovulation | 91 (12) | 121 (19)
  Treatment month 1 luteal: number analyzed (Participants) | 43 | 33
  Treatment month 1 luteal | 126 (11) | 108 (12)
  Treatment month 2 follicular: number analyzed (Participants) | 39 | 32
  Treatment month 2 follicular | 40 (6) | 35 (3)
  Treatment month 2 ovulation: number analyzed (Participants) | 21 | 14
  Treatment month 2 ovulation | 122 (19) | 113 (13)
  Treatment month 2 luteal: number analyzed (Participants) | 35 | 28
  Treatment month 2 luteal | 112 (9) | 101 (10)
Statistical Analysis 1: Comparison: Fluoxetine vs Bupropion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.4, Mixed Models Analysis
Statistical Analysis 2: Comparison: Fluoxetine vs Bupropion; This secondary analysis examined main effect of menstrual cycle phase on hormone levels; Test type: Superiority or Other; p < .0001, Mixed Models Analysis

5. Secondary Outcome: Change in Prolactin
Description: Hormone levels at early follicular, ovulation, and luteal phase of 3 menstrual cycles which included baseline month, month 1 of daily antidepressant treatment and month 2 of daily antidepressant treatment. Differential effects of the two antidepressant treatments and menstrual cycle on hormone levels were examined.
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 45 | 38
ng/ml
  Baseline month follicular: number analyzed (Participants) | 44 | 38
  Baseline month follicular | 11.2 (0.7) | 11.0 (1.2)
  Baseline month ovulation: number analyzed (Participants) | 27 | 20
  Baseline month ovulation | 15.9 (1.7) | 14.1 (1.6)
  Baseline month luteal | 16.4 (1.4) | 15.4 (1.6)
  Treatment month 1 follicular: number analyzed (Participants) | 42 | 38
  Treatment month 1 follicular | 12.1 (1.1) | 11.7 (1.5)
  Treatment month 1 ovulation: number analyzed (Participants) | 24 | 18
  Treatment month 1 ovulation | 12.9 (1.4) | 16.0 (2.9)
  Treatment month 1 luteal: number analyzed (Participants) | 40 | 30
  Treatment month 1 luteal | 14.0 (1.4) | 16.6 (1.9)
  Treatment month 2 follicular: number analyzed (Participants) | 40 | 33
  Treatment month 2 follicular | 12.8 (1.0) | 10.8 (1.4)
  Treatment month 2 ovulation: number analyzed (Participants) | 21 | 14
  Treatment month 2 ovulation | 17.1 (3.3) | 18.3 (4.4)
  Treatment month 2 luteal: number analyzed (Participants) | 35 | 28
  Treatment month 2 luteal | 13.7 (1.0) | 12.1 (0.8)
Statistical Analysis 1: Comparison: Fluoxetine vs Bupropion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.7, Mixed Models Analysis
Statistical Analysis 2: Comparison: Fluoxetine vs Bupropion; This secondary analysis examined main effect of menstrual cycle phase on hormone levels; Test type: Superiority or Other; p < .0001, Mixed Models Analysis

6. Secondary Outcome: Change in Progesterone
Description: Hormone levels at early follicular, ovulation, and luteal phase of the cycle were averaged for the baseline pre-treatment month and compared to average values during the 1st and 2nd months of antidepressant treatment.
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 45 | 38
ng/ml
  Baseline month follicular: number analyzed (Participants) | 41 | 38
  Baseline month follicular | 0.66 (0.2) | 0.5 (0.4)
  Baseline month ovulation: number analyzed (Participants) | 26 | 20
  Baseline month ovulation | 2.4 (0.6) | 2.8 (0.9)
  Baseline month luteal | 9.5 (0.9) | 9.6 (1.1)
  Treatment month 1 follicular: number analyzed (Participants) | 41 | 38
  Treatment month 1 follicular | 0.7 (0.2) | 0.7 (0.2)
  Treatment month 1 ovulation: number analyzed (Participants) | 25 | 18
  Treatment month 1 ovulation | 2.4 (0.7) | 3.9 (1.2)
  Treatment month 1 luteal: number analyzed (Participants) | 43 | 33
  Treatment month 1 luteal | 8.4 (1.1) | 7.4 (1.0)
  Treatment month 2 follicular: number analyzed (Participants) | 38 | 33
  Treatment month 2 follicular | 0.6 (0.2) | 0.6 (0.08)
  Treatment month 2 ovulation: number analyzed (Participants) | 21 | 14
  Treatment month 2 ovulation | 2.9 (0.8) | 3.2 (1.2)
  Treatment month 2 luteal: number analyzed (Participants) | 35 | 28
  Treatment month 2 luteal | 8.6 (1.2) | 8.1 (1.2)
Statistical Analysis 1: Comparison: Fluoxetine vs Bupropion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.9, Mixed Models Analysis
Statistical Analysis 2: Comparison: Fluoxetine vs Bupropion; This secondary analysis examined main effect of menstrual cycle phase on hormone levels; Test type: Superiority or Other; p < .0001, Mixed Models Analysis

7. Secondary Outcome: Change in Dehydroepiandrosterone Sulfate (DHEA-S)
Description: as for outcome 5
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/ml
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 45 | 38
ug/ml
  Baseline month follicular: number analyzed (Participants) | 44 | 38
  Baseline month follicular | 1.6 (0.1) | 1.8 (0.1)
  Baseline month ovulation: number analyzed (Participants) | 27 | 20
  Baseline month ovulation | 1.8 (0.2) | 2.0 (0.2)
  Baseline month luteal | 1.6 (0.1) | 1.9 (.01)
  Treatment month 1 follicular: number analyzed (Participants) | 42 | 38
  Treatment month 1 follicular | 1.6 (0.1) | 1.9 (0.1)
  Treatment month 1 ovulation: number analyzed (Participants) | 22 | 17
  Treatment month 1 ovulation | 1.7 (0.2) | 1.9 (0.2)
  Treatment month 1 luteal: number analyzed (Participants) | 38 | 29
  Treatment month 1 luteal | 1.7 (0.2) | 1.9 (0.2)
  Treatment month 2 follicular: number analyzed (Participants) | 37 | 33
  Treatment month 2 follicular | 1.6 (0.2) | 1.8 (0.2)
  Treatment month 2 ovulation: number analyzed (Participants) | 20 | 14
  Treatment month 2 ovulation | 1.9 (0.3) | 1.8 (0.2)
  Treatment month 2 luteal: number analyzed (Participants) | 35 | 28
  Treatment month 2 luteal | 1.9 (0.2) | 1.9 (0.2)
Statistical Analysis 1: Comparison: Fluoxetine vs Bupropion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.9, Mixed Models Analysis
Statistical Analysis 2: Comparison: Fluoxetine vs Bupropion; This secondary analysis examined main effect of menstrual cycle phase on hormone levels; Test type: Superiority or Other; p > 0.9, Mixed Models Analysis

8. Secondary Outcome: Change in Androstenedione
Description: as for outcome 5
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 45 | 38
ng/ml
  Baseline month follicular: number analyzed (Participants) | 44 | 38
  Baseline month follicular | 0.84 (0.05) | 0.89 (0.05)
  Baseline month ovulation: number analyzed (Participants) | 27 | 18
  Baseline month ovulation | 1.13 (0.07) | 1.28 (0.10)
  Baseline month luteal: number analyzed (Participants) | 43 | 34
  Baseline month luteal | 1.31 (0.10) | 1.14 (0.07)
  Treatment month 1 follicular: number analyzed (Participants) | 42 | 38
  Treatment month 1 follicular | 0.89 (0.07) | 0.84 (0.06)
  Treatment month 1 ovulation: number analyzed (Participants) | 25 | 18
  Treatment month 1 ovulation | 1.13 (0.10) | 0.96 (0.06)
  Treatment month 1 luteal: number analyzed (Participants) | 43 | 33
  Treatment month 1 luteal | 1.04 (0.06) | 1.13 (0.08)
  Treatment month 2 follicular: number analyzed (Participants) | 40 | 33
  Treatment month 2 follicular | 0.79 (0.05) | .85 (.06)
  Treatment month 2 ovulation: number analyzed (Participants) | 21 | 14
  Treatment month 2 ovulation | 1.07 (0.12) | 1.00 (0.13)
  Treatment month 2 luteal: number analyzed (Participants) | 34 | 28
  Treatment month 2 luteal | 1.13 (0.09) | 1.12 (0.12)
Statistical Analysis 1: Comparison: Fluoxetine vs Bupropion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.1, Mixed Models Analysis
Statistical Analysis 2: Comparison: Fluoxetine vs Bupropion; This secondary analysis examined main effect of menstrual cycle phase on hormone levels; Test type: Superiority or Other; p > 0.7, Mixed Models Analysis

9. Secondary Outcome: C-reactive Protein
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: This measure was not performed due to lack of anticipated supplementary funding.
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Inflammatory Cytokines
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: This measure was not performed due to lack of anticipated supplementary funding.
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Lymphocyte Activation Markers
Time Frame: Measured in baseline menstrual cycle and during antidepressant treatment for two menstrual cycles
Population: This measure was not performed due to lack of anticipated supplementary funding.
Arm/Group | Fluoxetine | Bupropion
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Each subject was assessed for 3 months.
Arm/Group | Fluoxetine | Bupropion
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/45 | 2/38
Other Adverse Events (participants affected / at risk) | 33/45 | 21/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluoxetine (N=45) | Bupropion (N=38)
seizure (Nervous system disorders) | 0 | 1
pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=45) | Bupropion (N=38)
reduced orgasm (Reproductive system and breast disorders) | 10 (10) | 6 (6)
reduced libido (Reproductive system and breast disorders) | 9 (9) | 3 (3)
reduced appetite (Gastrointestinal disorders) | 9 (9) | 11 (11)
dry mouth (Gastrointestinal disorders) | 5 (5) | 10 (10)
anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
yawning (Nervous system disorders) | 8 (8) | 4 (4)
diarrhea (Gastrointestinal disorders) | 6 (6) | 5 (5)
fatigue (General disorders) | 11 (11) | 7 (7)
headache (Nervous system disorders) | 14 (14) | 6 (6)
nausea (Gastrointestinal disorders) | 9 (9) | 12 (12)
insomnia (General disorders) | 6 (6) | 4 (4)
tinnitus (Nervous system disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes